CLINICAL TRIAL: NCT07136142
Title: A Multicenter, Open Label Phase I/II Clinical Study on the Safety, Tolerability, Pharmacokinetics and Efficacy of FH-006 for Injection in Patients With Malignant Solid Tumors
Brief Title: A Phase I/II Clinical Study of FH-006 for Injection in Patients With Malignant Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FH-006-102
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Malignant Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FH-006 Group (Experimental): FH-006 for injection monotherapy should be conducted.
  Interventions: Drug: FH-006 for Injection

INTERVENTIONS:
Drug: FH-006 for Injection — FH-006 for injection.

SUMMARY:
This study aims to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of FH-006 in subjects with advanced malignant solid tumors, and determine the preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with ability to understand and voluntarily agree to participate by giving written informed consent for the study.
2. Patients with unresectable recurrent or metastatic solid tumors.
3. There is at least one lesion that could be measured.
4. An Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1.
5. Adequate organ functions as defined.
6. Life expectancy ≥ 3 months.

Exclusion Criteria:

1. Patients with known active central nervous system (CNS) metastases.
2. Subjects who had other malignancy in five years before the first dose.
3. Patients with tumor-related pain that can not be controlled as determined.
4. Patients with serious cardiovascular and cerebrovascular diseases.
5. Uncontrollable third-space effusion, such as pleural effusion, pericardial effusion or peritoneal effusion.
6. Patients with severe infections.
7. History of immunodeficiency.
8. History of autoimmune diseases.
9. Unresolved CTCAE Grade >1 toxicity attributed to any prior anti-tumor therapy.
10. Active infection.
11. Pregnant or nursing women.
12. Known history of serious allergic reactions to the investigational product or its main ingredients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Assessed up to 6 months.
  ORR is the efficacy endpoint of FH-006 for injection monotherapy in treatment of patients with advanced solid tumors.

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | Up to 2 years.
Maximum concentration (Cmax) | Up to 2 years.
Terminal half-life (t1/2) | Up to 2 years.
Area Under the Concentration Versus Time Curve From Time Zero to T (AUC0-t) | Up to 2 years.
Adverse events (AEs) | Up to 24 weeks.
Serious adverse events (SAEs) | Up to 24 weeks.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Tianjin Medical Unversity Cancer Institute & Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided